CLINICAL TRIAL: NCT02454218
Title: Effect of Transcranial Direct-current Stimulation in Attentional Performance and Pain in Patients With Fibromyalgia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 140231
Record Dates: First submitted 2015-01-19; First posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Transcranial direct current stimulation
MeSH Terms: conditions — Fibromyalgia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Direct Current Stimulation (Active Comparator): The intensity of the asset is little perceived and painless.
  Interventions: Device: Transcranial Direct Current Stimulation
- Simulation Transcranial Current (Placebo Comparator): Will receive only simulation.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — The intervention session with tDCS lasts for 20 minutes. tDCS uses rubber electrodes that are within sponges that are moistened with saline. These electrodes are placed on the participant's head. Through these electrodes will pass a weak electrical current that can at most cause mild itching at the site where the electrode is positioned. The generated electric current is equivalent to a small common battery that we use to run toys or radios. The procedure does not require that the patient be subjected to shocks, cuts or surgery.
  The participant will receive active tDCS or placebo, but receive both types of intervention during the performance of the two sessions.
  Other Names: tDCS -

SUMMARY:
tDCS can modify the attentional response of patients with fibromyalgia. Methods: This study deals with a randomized, blind, crossover, controlled tDCS-sham. The sample will consist of 40 patients, divided into two groups with sham interventions and active crossover.

DETAILED DESCRIPTION:
Check that the tDCS can modify the attentional response of patients with fibromyalgia. Methods: This study deals with a randomized, blind, crossover, controlled tDCS-sham. The sample will consist of 40 patients, divided into two groups with sham interventions and active crossover. Patients answer the questionnaires in order to verify the Psychological Factors and Clinical. Will use the Impact of Fibromyalgia (QIF), Pittsburgh Sleep Questionnaire, Conditioned Pain Modulation (CPM), Beck Depression Scale II, Catastrophic Scale , Go noGo Test, Attention Network Task (ANT) to verify the ability attentional as well as to verify the Near-infrared spectroscopy (NIRS) brain oxygenation. They will be used before, during and after the intervention with tDCS. Intervention with tDCS or sham will be held in a single session. Expected results: It is expected that fibromyalgia patients undergoing tDCS present, after the intervention, improved attention capacity .

ELIGIBILITY:
Inclusion Criteria:

* Female patients, literate, right-handed, 18 to 65 years of age, who meet the criteria of the American College of Rheumatology (ACR) for fibromyalgia.

Exclusion Criteria:

* Pregnant women
* Contraindications to tDCS
* Metal implant in the brain
* History of alcohol or drug abuse in the last six months
* Suffer from severe depression (score> 30 on the Beck Depression Inventory)
* History of neurological disorders
* Unexplained fainting
* Self-reports of head injury or momentary loss of awareness
* Neurosurgery.
* Will also be excluded patients who have decompensated systemic diseases and / or chronic inflammatory diseases (ex .: lupus, rheumatoid arthritis).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-05 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Attention capacity after the intervention, assessed by the Attention Network Task | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei M Caumo, M.D., PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Porto Alegre Clinical Hospital, Porto Alegre, Rio Grande do Sul, Brazil